CLINICAL TRIAL: NCT04142489
Title: Clinical Study of In Vivo Damage Induced bu UV in the Epidermis of the Scalp
Brief Title: In Vivo Damage Induced bu UV in the Epidermis of the Scalp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-AOIP-02
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Squamous Cell Carcinomas
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UV and biopsy (Other): Minimum erythematous dose (DEM) will be calculated using a solar irradiator on the scalp (study area) and on a forearm (control area). On D2 (D1+24h) a solar irradiation corresponding to 2 DEM will be performed on a region of the scalp (studied area), as well as on a forearm (control area). A 3mm biopsy will be performed 15mn after irradiation in these 2 regions to study DNA damage. At D4 (D2+48h) a 2nd biopsy of 3 mm will be performed to study the repair of induced DNA damage. The study of DNA damage induced by UV will be done by immunohistochemical analysis of markers validated in previous studies: CPD=pyridine dimers, 6.4 PP= "6.4 photoproducts", and p53. Immunolabeling will be performed on skin biopsies collected 15 minutes after UV exposure and 48 hours after UV exposure.
  Interventions: Other: solar irradiation and biopsies

INTERVENTIONS:
Other: solar irradiation and biopsies — the minimum erythematous dose (DEM) will be calculated using a solar irradiator on the scalp (study area) and on a forearm (control area). On D2 (D1+24h) a solar irradiation corresponding to 2 DEM will be performed on a region of the scalp (studied area), as well as on a forearm (control area). A 3mm biopsy will be performed 15mn after irradiation in these 2 regions to study DNA damage. At D4 (D2+48h) a 2nd biopsy of 3 mm will be performed to study the repair of induced DNA damage.

SUMMARY:
Squamous cell carcinomas (SCC) are the second most common skin cancer in humans. The incidence of SCCs in the USA in 2012 was estimated at 700,000 casesSCCs have a metastatic course in 3% to 5% of cases that is of poor prognosis. In men, the SCCs of the scalp represent the most frequent location of the head and neck, the 3rd location of the whole body. The SCCs of the scalp are more undifferentiated than in other locations. In addition, actinic keratoses of scalp, precursors of SCC, are more resistant to treatment than in other areas. These particularities of the SCCs of the scalp suggest the existence of specific factors at the epidermis level of the scalp.

UV-induced damage to DNA is the defining event in skin photocarcinogenesis. It has already been shown that DNA damage induced by UV and the kinetics of repair of this damage may vary with age or phototype of patients, but the topographic variation of DNA damage has never been studied, although it is known that gene expression in skin cells may differ from one region of the body to another.

the hypothesis is therefore that the particular characteristics of KAs and SCCs at the scal level could be explained by an increased sensitivity to UV-induced damage. It is planned to study UV-induced damage and its repair at the scalp level in humans compared to the forearm.

ELIGIBILITY:
Inclusion Criteria:

* Male subject
* Subject aged 40 to 60 years
* Subject of phototype III or IV
* Subject with no skin lesions on the scalp and forearms
* Subject who has not been exposed to the sun for at least 1 month
* Subject affiliated to social security
* Subject who signed the informed consent form

Exclusion Criteria:

* Subjects with photosensitivity,
* Subject taking photosensitizing drugs
* Subjects with a history of skin cancer
* Subjects with abnormal healing
* Subjects with immunosuppression

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
number oh epidermal cells positives | 6 months
  epidermal cells with positive immunolabeling for DNA damage markers (CPD, 6.4PP, p53) count.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No